CLINICAL TRIAL: NCT00698022
Title: A 4-week, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Mifepristone in the Prevention of Risperidone-induced Weight Gain in Healthy Male Volunteers
Brief Title: A 4-week Study of Mifepristone in the Prevention of Risperidone-induced Weight Gain in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: C-1073-205
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: healthy; weight gain; anti-psychotic; risperidone; mifepristone; mitigation; weight loss
MeSH Terms: conditions — Weight Gain; Weight Loss | interventions — Risperidone; Mifepristone; Corlux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Risperidone plus mifepristone (Experimental): risperidone plus mifepristone daily for 28 days
  Interventions: Drug: Risperidone; Drug: Mifepristone
- Risperidone plus mifepristone-matched placebo (Placebo Comparator): risperidone plus mifepristone-matched placebo daily for 28 days
  Interventions: Drug: Risperidone; Drug: Mifepristone-matched placebo
- Risperidone-matched placebo plus mifepristone (Placebo Comparator): risperidone-matched placebo plus mifepristone daily for 28 days
  Interventions: Drug: Mifepristone; Drug: Risperidone-matched placebo

INTERVENTIONS:
Drug: Risperidone — risperidone daily for 28 days
  Other Names: Risperdal
  Arms: Risperidone plus mifepristone; Risperidone plus mifepristone-matched placebo
Drug: Mifepristone — mifepristone daily for 28 days
  Other Names: Corlux
  Arms: Risperidone plus mifepristone; Risperidone-matched placebo plus mifepristone
Drug: Risperidone-matched placebo — risperidone-matched placebo daily for 28 days
  Arms: Risperidone-matched placebo plus mifepristone
Drug: Mifepristone-matched placebo — mifepristone-matched placebo daily for 28 days
  Arms: Risperidone plus mifepristone-matched placebo

SUMMARY:
This is a 28-day, single-center, double-blind, placebo-controlled inpatient study of the administration of risperidone alone or in combination with mifepristone in healthy adult male volunteers to determine the average change in absolute weight at Day 28 compared to baseline.

DETAILED DESCRIPTION:
This is a 28-day, single-center, double-blind, placebo-controlled inpatient study of the administration of risperidone alone or in combination with mifepristone in healthy adult male volunteers. The primary study objective is to determine the mean change in absolute weight at Day 28 compared to baseline in normal healthy male volunteers treated with risperidone plus mifepristone or risperidone alone. The secondary study objectives are to determine the mean percent change in baseline body weight; and the proportion of subjects that gain less than 5% and less than 7% of their baseline body in the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18 and ≤ 23 kg/m2
* Able to provide written informed consent
* Routine clinical laboratory tests either within normal limits or not clinically meaningful if outside of normal limits
* AST, ALT, Tbili within normal limits at screening
* Medical and psychiatric history and physical examination devoid of any significant findings that would interfere with participation or interpretation of results in this study
* Agree to use a barrier method of birth control for 28 days following the last dose of study medication
* Have maintained a stable weight for at least 6 months prior to Screening

Exclusion Criteria:

* Prior or current history of any psychiatric disorder, including eating disorders such as anorexia nervosa, bulimia nervosa, or binge-eating disorder
* Positive urine drug screen for any drug of abuse (including amphetamines, cannabinoids, barbiturates, cocaine, opiates, benzodiazepines) unless prescribed by a physician
* Participation in a clinical investigation of any drug, biological or other investigational therapy within 30 days prior to dosing
* Have a history of an allergic reaction to either mifepristone or risperidone
* Any other clinically significant abnormality on screening laboratory tests
* QTc Bazzett's ≥ 450 msec
* History of or current major medical condition, which in the opinion of the Investigator would place the patient at undue risk.
* Receiving any prescription or over-the-counter medications that could potentially affect appetite or weight
* Any history of a movement disorder such as Tardive Dyskinesia, Parkinsonism
* Any personal or family history of Neuroleptic Malignant Syndrome

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleman Gross, MD, Study Director — Corcept Therapeutics
Locations (1):
- Dhirubhai Ambani Life Sciences Centre, Mumbai, India

REFERENCES:
- [Background] Beebe KL, Block T, Debattista C, Blasey C, Belanoff JK. The efficacy of mifepristone in the reduction and prevention of olanzapine-induced weight gain in rats. Behav Brain Res. 2006 Aug 10;171(2):225-9. doi: 10.1016/j.bbr.2006.03.039. Epub 2006 Jun 19. PMID 16782211
- See also: Sponsor's Website — http://www.corcept.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone Plus Risperidone: mifepristone plus risperidone daily
- Risperidone Plus Mifepristone-matched Placebo: risperidone plus mifepristone-matched placebo daily
- Risperidone-matched Placebo Plus Mifepristone: risperidone-matched placebo plus mifepristone daily
Period: Overall Study
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
Started | 30 | 30 | 16
Completed | 14 | 20 | 14
Not Completed | 16 | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone | Total
Number analyzed (Participants) | 30 | 30 | 16 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 16 | 76
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.9) | 25.6 (3.6) | 24.9 (4.6) | 25 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 30 | 16 | 76
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 16 | 76
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 57.5 (4.1) | 60.4 (4.7) | 58.2 (4.1) | 58.8 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline and 28 days
Population: All randomized participants who had at least one post baseline assessment.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
Number analyzed (Participants) | 30 | 30 | 16
kilograms | 2.32 (0.32) | 4.23 (0.33) | 2.87 (0.43)

2. Secondary Outcome: Percentage of Participants With <5% and <7% Increase From Baseline in Body Weight
Time Frame: Baseline and 28 days
Population: All participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
Number analyzed (Participants) | 14 | 20 | 14
Participants
  <5% increase in body weight | 9 | 3 | 8
  <7% increase in body weight | 13 | 10 | 11

3. Secondary Outcome: Percentage of Participants With One or More Adverse Events
Time Frame: Up to 28 days
Population: All participants who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
Number analyzed (Participants) | 30 | 30 | 16
Participants | 29 | 27 | 13

4. Secondary Outcome: Percentage of Participants Discontinued From the Study Due to an Adverse Event
Time Frame: Up to 28 days
Population: All participants who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
Number analyzed (Participants) | 30 | 30 | 16
Participants | 5 | 4 | 1

ADVERSE EVENTS:
Arm/Group | Mifepristone Plus Risperidone | Risperidone Plus Mifepristone-matched Placebo | Risperidone-matched Placebo Plus Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 1/16
Other Adverse Events (participants affected / at risk) | 2/30 | 3/30 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone Plus Risperidone (N=30) | Risperidone Plus Mifepristone-matched Placebo (N=30) | Risperidone-matched Placebo Plus Mifepristone (N=16)
suspected snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mifepristone Plus Risperidone (N=30) | Risperidone Plus Mifepristone-matched Placebo (N=30) | Risperidone-matched Placebo Plus Mifepristone (N=16)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days